CLINICAL TRIAL: NCT06009991
Title: The Investigation of the Dose Range of Remimazolam Besylate in Different Age Groups of Adults and Its Effects on Hemodynamics
Brief Title: The Dose Range of Remimazolam Besylate in Different Age Groups
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Renmin Hospital of Wuhan University (Other); Wuhan University (Other); The General Hospital of Central Theater Command (Other); Taihe Hospital (Other); Yichang Central People's Hospital (Other); Jingzhou Central Hospital (Other); Beijing Shijitan Hospital, Capital Medical University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); First Affiliated Hospital of Fujian Medical University (Other); Tianjin Nankai Hospital (Other); Sichuan Provincial People's Hospital (Other); Shanxi Bethune Hospital (Other)
Responsible Party: Principal Investigator, Ailin Luo, Professor and Chief Physician, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TongjiHospital-Anes QQ02
Record Dates: First submitted 2023-08-17; First posted 2023-08-24 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Remimazolam; Anesthesia
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Age 45-64 (Experimental): Patients aged 45 to 64 years
  Interventions: Drug: Remimazolam besylate; Drug: Propofol
- Age 65-74 (Experimental): Patients aged 65 to 74 years
  Interventions: Drug: Remimazolam besylate; Drug: Propofol
- Age 75-84 (Experimental): Patients aged 75 to 84 years
  Interventions: Drug: Remimazolam besylate; Drug: Propofol
- Age over 75 (Experimental): Patients aged over 85 years
  Interventions: Drug: Remimazolam besylate; Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam besylate — Age 45-64: Remimazolam Besylate 0.3 mg/kg for anesthesia induction (0.05mg/kg for additional need) and 0.5mg/kg/h for maintenance (0.25 mg/kg/h for additional need).
  Age over 65: Remimazolam Besylate 0.15 mg/kg for anesthesia induction (0.05mg/kg for additional need) and 0.5mg/kg/h for maintenance (0.25 mg/kg/h for additional need).
Drug: Propofol — Age 45-64: Propofol 3.0μg/ml TCI for anesthesia induction and 2.5-3.0μg/ml TCI for maintenance.
  Age over 65: Propofol 1.5-2.5μg/ml TCI for anesthesia induction and 1.5-2.5μg/ml TCI for maintenance

SUMMARY:
This is a multicenter, randomized, parallel, controlled clinical study of patients at different ages underwent elective non-cardiac surgery under general anesthesia. The aim of this study is to explore the dose range of remimazolam besylate for patients at different ages, to provide guidance for anesthesia induction and maintenance of remimazolam besylate. And to investigate the incidence of perioperative hypotension and postoperative related organ dysfunction in patients received total intravenous anesthesia with remimazolam besylate, compared with propofol.

DETAILED DESCRIPTION:
Surgery is an effective method to treat surgical diseases, prolong survival time and improve the quality of life, but patients often face the risk of postoperative complications. In general surgery patients, complications occur in more than 30% of patients. Several observational studies have shown that the severity and duration of intraoperative hypotension are significantly related to the risk of postoperative adverse events such as myocardial injury, renal injury, stroke, delirium, prolonged hospitalization, and death.

Hypotension, defined as a systolic blood pressure of less than 90 mmHg, a diastolic blood pressure of less than 50 mmHg, or a 20% reduction in systolic blood pressure from baseline, is common during anesthesia and surgery. More than a third of patients receiving propofol sedation experience intraoperative hypotension events, and their duration and degree are associated with harm during surgery.

Remimazolam is a new ultra-short-acting sedative drug developed in recent years, which has a similar structure to midazolam. However, compared with midazolam, remimazolam has the advantages of faster onset, faster recovery, and higher safety. Compared with propofol, remimazolam is noninferior in the success rate of sedation, while the incidence of adverse events such as hypotension is lower. At present, remimazolam has completed phase III clinical studies in many fields, such as colonoscopy, fiberoptic bronchoscopy, and general anesthesia induction and maintenance, which have shown its safety and effectiveness. However, there may be differences in hemodynamics and drug sensitivity among patients of different ages. Compared with young patients, elderly patients have a higher risk of hypotension after anesthesia induction. At present, there is a lack of clinical studies with large samples to clarify the recommended dose of remimazolam for anesthesia induction and maintenance in patients of all ages. The updated instructions for remimazolam besylate for injection on March 28, 2022 also mention that remimazolam besylate is used as a sedative drug for general anesthesia induction and maintenance, and the relevant dose reference is given. However, the safety and effectiveness of patients over 65 years have not been confirmed. The precise regulation of clinical use for patients of different ages and the optimization of drug dosage during anesthesia induction and maintenance are the basis for ensuring the safety of clinical medication at present., in order to maintain the stability of perioperative hemodynamics, and prevent or reduce the occurrence of adverse cardiovascular events.

This study aims to investigate the effect of remimazolam total intravenous anesthesia on intraoperative hemodynamics and the drug requirement for patients of different ages, with propofol as the control, and intraoperative hemodynamics as the main evaluation index, so as to provide evidence for clinical application of remimazolam for elderly patients in anesthesia induction and maintenance.

ELIGIBILITY:
Inclusion Criteria:

1. age above 45 years old;
2. American Society of Anesthesiologists grade Ⅰ-II;
3. patients undergoing tracheal intubation or laryngeal mask airway surgery under general anesthesia (intravenous anesthesia);
4. Informed consent: patients voluntarily participated in the trial and signed the informed consent form.

Exclusion Criteria:

1. patients with cardiac function grade 3 or above;
2. difficult to observe the pupil size of head or neck surgery patients;
3. patients with multimodal anesthesia such as nerve block or spinal anesthesia compounded;
4. patients known to be allergic to remimazolam besylate or benzodiazepines;
5. major vascular surgery and the type of surgery that directly affects hemodynamics;
6. patients with coagulation dysfunction, endocrine diseases or other hemodynamic conditions;
7. minor surgery (operation duration <1 hour);
8. surgery lasting more than 4 hours;
9. emergency surgery;
10. patients with a history of drug or alcohol dependence;
11. Subjects deemed unsuitable for the study by the investigator.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1876 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of intraoperative hypotension | Operation 1 day
  Occurrence of intraoperative hypotension

SECONDARY OUTCOMES:
Intraoperative dosage of vasoactive drugs | Operation 1 day
  Intraoperative dosage of vasoactive drugs
Anesthesia recovery | Operation 1 day
  Anesthesia recovery
Cognitive function assessment | Operation 1 day
  Cognitive function assessment in the anesthesia recovery room
Major organ complications | Within 30 days after surgery
  The occurrence of major organ complications within 30 days after surgery
Hospital stay of patients | With 30 days after surgery
  Hospital stay of patients
30-day mortality after surgery | 30-day after surgery
  30-day mortality after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ailin Luo, Principal Investigator — Tongji Hospital
Locations (1):
- ongji Hospital, Tongji Medical College, Huazhong Science and Technology University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
This is a multicenter clinical study and the plan need depend on multiple hospital views.

REFERENCES:
- [Result] Ghaferi AA, Birkmeyer JD, Dimick JB. Complications, failure to rescue, and mortality with major inpatient surgery in medicare patients. Ann Surg. 2009 Dec;250(6):1029-34. doi: 10.1097/sla.0b013e3181bef697. PMID 19953723
- [Result] Wesselink EM, Kappen TH, Torn HM, Slooter AJC, van Klei WA. Intraoperative hypotension and the risk of postoperative adverse outcomes: a systematic review. Br J Anaesth. 2018 Oct;121(4):706-721. doi: 10.1016/j.bja.2018.04.036. Epub 2018 Jun 20. PMID 30236233
- [Result] Mascha EJ, Yang D, Weiss S, Sessler DI. Intraoperative Mean Arterial Pressure Variability and 30-day Mortality in Patients Having Noncardiac Surgery. Anesthesiology. 2015 Jul;123(1):79-91. doi: 10.1097/ALN.0000000000000686. PMID 25929547
- [Result] Salmasi V, Maheshwari K, Yang D, Mascha EJ, Singh A, Sessler DI, Kurz A. Relationship between Intraoperative Hypotension, Defined by Either Reduction from Baseline or Absolute Thresholds, and Acute Kidney and Myocardial Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2017 Jan;126(1):47-65. doi: 10.1097/ALN.0000000000001432. PMID 27792044
- [Result] Babazade R, Yilmaz HO, Zimmerman NM, Stocchi L, Gorgun E, Kessler H, Sessler DI, Kurz A, Turan A. Association Between Intraoperative Low Blood Pressure and Development of Surgical Site Infection After Colorectal Surgery: A Retrospective Cohort Study. Ann Surg. 2016 Dec;264(6):1058-1064. doi: 10.1097/SLA.0000000000001607. PMID 26756765
- [Result] Futier E, Lefrant JY, Guinot PG, Godet T, Lorne E, Cuvillon P, Bertran S, Leone M, Pastene B, Piriou V, Molliex S, Albanese J, Julia JM, Tavernier B, Imhoff E, Bazin JE, Constantin JM, Pereira B, Jaber S; INPRESS Study Group. Effect of Individualized vs Standard Blood Pressure Management Strategies on Postoperative Organ Dysfunction Among High-Risk Patients Undergoing Major Surgery: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1346-1357. doi: 10.1001/jama.2017.14172. PMID 28973220
- [Result] Hallqvist L, Granath F, Fored M, Bell M. Intraoperative Hypotension and Myocardial Infarction Development Among High-Risk Patients Undergoing Noncardiac Surgery: A Nested Case-Control Study. Anesth Analg. 2021 Jul 1;133(1):6-15. doi: 10.1213/ANE.0000000000005391. PMID 33555690
- [Result] Ahuja S, Mascha EJ, Yang D, Maheshwari K, Cohen B, Khanna AK, Ruetzler K, Turan A, Sessler DI. Associations of Intraoperative Radial Arterial Systolic, Diastolic, Mean, and Pulse Pressures with Myocardial and Acute Kidney Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2020 Feb;132(2):291-306. doi: 10.1097/ALN.0000000000003048. PMID 31939844
- [Result] Sneyd JR, Absalom AR, Barends CRM, Jones JB. Hypotension during propofol sedation for colonoscopy: a retrospective exploratory analysis and meta-analysis. Br J Anaesth. 2022 Apr;128(4):610-622. doi: 10.1016/j.bja.2021.10.044. Epub 2021 Dec 13. PMID 34916051
- [Result] Chen SH, Yuan TM, Zhang J, Bai H, Tian M, Pan CX, Bao HG, Jin XJ, Ji FH, Zhong TD, Wang Q, Lv JR, Wang S, Li YJ, Yu YH, Luo AL, Li XK, Min S, Li L, Zou XH, Huang YG. Remimazolam tosilate in upper gastrointestinal endoscopy: A multicenter, randomized, non-inferiority, phase III trial. J Gastroenterol Hepatol. 2021 Feb;36(2):474-481. doi: 10.1111/jgh.15188. Epub 2020 Jul 24. PMID 32677707
- [Result] Rex DK, Bhandari R, Desta T, DeMicco MP, Schaeffer C, Etzkorn K, Barish CF, Pruitt R, Cash BD, Quirk D, Tiongco F, Sullivan S, Bernstein D. A phase III study evaluating the efficacy and safety of remimazolam (CNS 7056) compared with placebo and midazolam in patients undergoing colonoscopy. Gastrointest Endosc. 2018 Sep;88(3):427-437.e6. doi: 10.1016/j.gie.2018.04.2351. Epub 2018 Apr 30. PMID 29723512
- [Result] Pastis NJ, Yarmus LB, Schippers F, Ostroff R, Chen A, Akulian J, Wahidi M, Shojaee S, Tanner NT, Callahan SP, Feldman G, Lorch DG Jr, Ndukwu I, Pritchett MA, Silvestri GA; PAION Investigators. Safety and Efficacy of Remimazolam Compared With Placebo and Midazolam for Moderate Sedation During Bronchoscopy. Chest. 2019 Jan;155(1):137-146. doi: 10.1016/j.chest.2018.09.015. Epub 2018 Oct 4. PMID 30292760
- [Result] Doi M, Morita K, Takeda J, Sakamoto A, Yamakage M, Suzuki T. Efficacy and safety of remimazolam versus propofol for general anesthesia: a multicenter, single-blind, randomized, parallel-group, phase IIb/III trial. J Anesth. 2020 Aug;34(4):543-553. doi: 10.1007/s00540-020-02788-6. Epub 2020 May 16. PMID 32417976
- [Result] Doi M, Hirata N, Suzuki T, Morisaki H, Morimatsu H, Sakamoto A. Safety and efficacy of remimazolam in induction and maintenance of general anesthesia in high-risk surgical patients (ASA Class III): results of a multicenter, randomized, double-blind, parallel-group comparative trial. J Anesth. 2020 Aug;34(4):491-501. doi: 10.1007/s00540-020-02776-w. Epub 2020 Apr 17. PMID 32303884
- [Result] Chen B, Pang QY, An R, Liu HL. A systematic review of risk factors for postinduction hypotension in surgical patients undergoing general anesthesia. Eur Rev Med Pharmacol Sci. 2021 Nov;25(22):7044-7050. doi: 10.26355/eurrev_202111_27255. PMID 34859868
- [Result] Saugel B, Reese PC, Sessler DI, Burfeindt C, Nicklas JY, Pinnschmidt HO, Reuter DA, Sudfeld S. Automated Ambulatory Blood Pressure Measurements and Intraoperative Hypotension in Patients Having Noncardiac Surgery with General Anesthesia: A Prospective Observational Study. Anesthesiology. 2019 Jul;131(1):74-83. doi: 10.1097/ALN.0000000000002703. PMID 30998509
- [Result] Ard JL, Kendale S. Searching for baseline blood pressure: A comparison of blood pressure at three different care points. J Clin Neurosci. 2016 Dec;34:59-62. doi: 10.1016/j.jocn.2016.08.001. Epub 2016 Aug 17. PMID 27544232
- [Result] Mathis MR, Naik BI, Freundlich RE, Shanks AM, Heung M, Kim M, Burns ML, Colquhoun DA, Rangrass G, Janda A, Engoren MC, Saager L, Tremper KK, Kheterpal S, Aziz MF, Coffman T, Durieux ME, Levy WJ, Schonberger RB, Soto R, Wilczak J, Berman MF, Berris J, Biggs DA, Coles P, Craft RM, Cummings KC, Ellis TA 2nd, Fleishut PM, Helsten DL, Jameson LC, van Klei WA, Kooij F, LaGorio J, Lins S, Miller SA, Molina S, Nair B, Paganelli WC, Peterson W, Tom S, Wanderer JP, Wedeven C; Multicenter Perioperative Outcomes Group Investigators. Preoperative Risk and the Association between Hypotension and Postoperative Acute Kidney Injury. Anesthesiology. 2020 Mar;132(3):461-475. doi: 10.1097/ALN.0000000000003063. PMID 31794513